CLINICAL TRIAL: NCT00904215
Title: A Post Marketing Observational Study to Investigate the Efficacy, Safety, Tolerability and the Effect on Quality of Life of Telmisartan (Micardis) and Telmisartan With HCTZ (Micardis Plus) in Patients With Hypertension
Brief Title: An Observational Study to Investigate the Efficacy, Safety, Tolerability and the Effect on Quality of Life of Telmisartan (Micardis) and Telmisartan With HCTZ (Micardis Plus) in Patients With Hypertension
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Other Study IDs: 502.487
Record Dates: First submitted 2009-05-18; First posted 2009-05-19 (Estimated); Results first posted 2009-08-31 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-04

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Telmisartan; Hydrochlorothiazide

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Drug: telmisartan/telmisartan + HCTZ (Hydrochlorothiazide)

SUMMARY:
An observational study to investigate the efficacy, safety, tolerability and the effect on quality of life of Telmisartan (Micardis) and Telmisartan with HCTZ (Micardis Plus) in patients with hypertension

ELIGIBILITY:
Inclusion Criteria:

1. Ability to provide written/verbal informed consent in accordance with GCP (Good Clinical Practice) and local legislation
2. Patients aged 18 ~ under 80
3. Hypertension as described below:

   * Newly diagnosed patients with hypertension
   * Patients with current antihypertensive therapy

Exclusion Criteria:

1. Female subjects who are breastfeeding, pregnant or who plan to be pregnant during the study
2. Known or suspected secondary hypertension(e.g. pheochromocytoma)
3. Patients who have been treated with telmisartan prior to the acquisition of informed consent (including verbal informed consent)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from clinics and hospitals in Korea
Sampling Method: Probability Sample
Enrollment: 1095 (Actual)
Dates: Start 2005-02; Primary Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (11):
- South Korea (11):
  - Boehringer ingelheim Investigational Site 1, Daegu
  - Boehringer ingelheim Investigational Site 4, Daegu
  - Boehringer ingelheim Investigational Site 7, Daegu
  - Boehringer ingelheim Investigational Site 9, Daejeon
  - Boehringer ingelheim Investigational Site 10, Koyang
  - Boehringer ingelheim Investigational Site 11, Kwangju
  - Boehringer ingelheim Investigational Site 3, Kwangju
  - Boehringer ingelheim Investigational Site 5, Pusan
  - Boehringer ingelheim Investigational Site 2, Seoul
  - Boehringer ingelheim Investigational Site 6, Suwon
  - Boehringer ingelheim Investigational Site 8, Wŏnju

RESULTS

PARTICIPANT FLOW:
Groups:
- Micardis/Micardis Plus: Patients aged 18~80 with hypertension who took Micardis/Micardis Plus
Period: Overall Study
Arm/Group | Micardis/Micardis Plus
Started | 1095
Completed | 960
Not Completed | 135
Not completed — Adverse Event | 25
Not completed — Protocol Violation | 10
Not completed — Lost to Follow-up | 63
Not completed — Withdrawal by Subject | 9
Not completed — Other | 28

BASELINE CHARACTERISTICS:
Arm/Group | Micardis/Micardis Plus
Number analyzed (Participants) | 1025
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 494
  Male | 531

OUTCOME MEASURES:

1. Primary Outcome: Change in SBP (Systolic Blood Pressure)
Description: The change of the mean SBP
Time Frame: between baseline (visit 1) and after 12 weeks of treatment (visit 3)
Population: In clinical report form (CRF), some patients' SBP was not recorded.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Micardis/Micardis Plus
Number analyzed (Participants) | 958
mmHg | -18 (19) [-19 to -17]
Statistical Analysis 1: Comparison: Micardis/Micardis Plus; Test type: Superiority or Other; p < 0.0001, Student Paired t-test

2. Primary Outcome: Change in DBP (Diastolic Blood Pressure)
Description: The change of the mean DBP
Time Frame: between baseline (visit 1) and after 12 weeks of treatment (visit 3)
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Micardis/Micardis Plus
Number analyzed (Participants) | 958
mmHg | -10 (12) [2.0 to 3.0]
Statistical Analysis 1: Comparison: Micardis/Micardis Plus; Test type: Superiority or Other; p < 0.0001, Student Paired t-test

3. Secondary Outcome: Change in VAS (Visual Analog Scale)
Description: VAS indicates the health status of the patient. Best value=100.0 (best health status), worst value=0.0 (worst health status)
Time Frame: between baseline (visit 1) and after 12 weeks of treatment (visit 3)
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Micardis/Micardis Plus
Number analyzed (Participants) | 918
Units on a scale | 5.9 (14.1) [5.0 to 6.9]
Statistical Analysis 1: Comparison: Micardis/Micardis Plus; Test type: Superiority or Other; p < 0.0001, Student Paired t-test

4. Primary Outcome: Change in WHO-QOL (WHO-Quality Of Life)
Description: World Health Organization-Quality Of Life (WHO-QOL), change in quality of life was assessed.
  Best value=130.0 (highest quality of life), worst value=0.0 (lowest quality of life)
Time Frame: between baseline (visit 1) and after 12 weeks of treatment (visit 3)
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Micardis/Micardis Plus
Number analyzed (Participants) | 956
Units on a scale | 2.5 (7.9) [2.0 to 3.0]
Statistical Analysis 1: Comparison: Micardis/Micardis Plus; Test type: Superiority or Other; p < 0.0001, Student Paired t-test

ADVERSE EVENTS:
Time Frame: After signing informed consent through the end of study
Arm/Group | Micardis/Micardis Plus
Serious Adverse Events (participants affected / at risk) | 8
Other Adverse Events (participants affected / at risk) | 0/1095
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Micardis/Micardis Plus
Cerebral infarction (Nervous system disorders) | 1/1095
Peritonitis (Gastrointestinal disorders) | 1/1095
Gastric polyps (Gastrointestinal disorders) | 1/1095
Gastric ulcer (Gastrointestinal disorders) | 1/1095
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1/1095
Varices oesophageal (Gastrointestinal disorders) | 1/1095
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1/1095
Hypertension (Vascular disorders) | 1/1095
Angina pectoris (Cardiac disorders) | 1/1095
Angina unstable (Cardiac disorders) | 1/1095
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/1095

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.